CLINICAL TRIAL: NCT07201324
Title: Analysis of the Relationships Between Cranial Remolding Orthosis Therapy, Cervical Spine Motor Function, and Thermoregulatory Responses in Children With Cranial Deformity
Brief Title: Effects of Corrective Helmet Therapy on Cervical Motion and Thermoregulation in Children With Positional Deformities
Status: Not yet recruiting | Type: Observational
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Natalia Zielińska, Master of Physiotherapy, Wroclaw University of Health and Sport Sciences
Other Study IDs: 26/2025
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Plagiocephaly, Nonsynostotic; Brachycephaly
Keywords: positional head deformity; helmet therapy; infants; thermoregulation; range of motion of the cervical spine
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic; Craniosynostoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cranial helmet therapy - observational — This observational study involves children undergoing cranial helmet therapy. The intervention is not assigned by the investigator. Repeated measurements are performed within participants to evaluate therapy effects. Stage 1 assesses head shape changes to analyze therapy effectiveness. Stage 2 examines factors influencing effectiveness, considering age, deformity type, and sex.
  Stage 3 measures body surface temperature using thermal imaging before, during, and after helmet use, with participants analyzed in three age groups: 4-6, 7-9, and 10-12 months. Stage 4 evaluates cervical spine rotation before therapy and after completion, with participants analyzed in the same three age groups.

SUMMARY:
The purpose of the study is to examine how cranial helmet therapy may affect neck movement and body temperature regulation in children with positional head deformity. The study will also look at factors that might influence how well the therapy works, such as the child's age, sex, and the type of head shape deformity.

During the study, children will undergo several assessments:

measurement of head shape using standard cranial indices, recording of body surface temperature with a thermal imaging camera, evaluation of neck mobility, focusing on rotation of the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* positional head deformity of severe or very severe degree;
* age at therapy initiation: 4-12 months;
* minimum therapy duration of 12 weeks (for Stage 1 and Stage 2).

Exclusion Criteria:

* craniosynostosis;
* hydrocephalus;
* non-adherence to 23-hour daily helmet use;
* metabolic disorders;
* torticollis.

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants are children from various cities in Poland, aged 4-12 months, diagnosed with severe or very severe positional head deformity and referred for cranial helmet therapy by a neurosurgeon. Both boys and girls are included. All referring physicians used the same standardized scale to determine the severity of the deformity, ensuring consistency across sites.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Cranial Index (CI) | Baseline (before therapy initiation) and after completion of cranial helmet therapy (average of 3-7 months after initiation).
  Assessment of cranial proportion using the Cranial Index (CI) in children undergoing cranial helmet therapy. Each participant serves as their own control.
Change in Cranial Vault Asymmetry Index (CVAI) | Baseline (before therapy initiation) and after completion of cranial helmet therapy (average of 3-7 months after initiation).
  Assessment of head shape asymmetry using the Cranial Vault Asymmetry Index (CVAI) in children undergoing cranial helmet therapy. Each participant serves as their own control.

SECONDARY OUTCOMES:
Factors Determining Therapy Effectiveness | Baseline (before therapy initiation) and after completion of cranial helmet therapy (average of 3-7 months after initiation)
  Analysis of how age, sex, and type of deformity influence changes in head shape. Same children as in Primary Outcome are included, divided according to age, deformity type, and sex.
Thermoregulatory Responses | Before helmet application, after 30 minutes of helmet use, immediately after removal, 10 minutes and 15 minutes post-removal
  Measurement of body surface temperature using thermal imaging to assess distribution and changes during and after cranial helmet therapy. Data will be analyzed in three age groups: 4-6, 7-9, and 10-12 months. Participants are different from those in the Primary Outcome.
Cervical Spine Rotation Range | Before therapy during helmet adaptation and after completion of cranial helmet therapy
  Assessment of neck rotation range in children to evaluate changes in cervical spine mobility. Measurements will be analyzed in three age groups: 4-6, 7-9, and 10-12 months.